CLINICAL TRIAL: NCT04992260
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase Ⅲ Clinical Trial to Evaluate the Efficacy, Immunogenicity and Safety of COVID-19 Vaccine(Vero Cell) ,Inactivated in Children and Adolescents Aged 6 Months to 17 Years
Brief Title: Efficacy, Immunogenicity and Safety of COVID-19 Vaccine , Inactivated in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-3002
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): subjects will receive two doses of inactivated COVID-19 vaccine on day 0 and day 28.
  Interventions: Biological: Inactivated COVID-19 Vaccine
- Control Group (Placebo Comparator): subjects will receive two doses of placebo on day 0 and day 28.
  Interventions: Biological: Controlled vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 Vaccine — The inactivated COVID-19 vaccine was manufactured by Sinovac Research& Development Co., Ltd..600SU Inactivated SARS-COV-2 virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Experimental Group
Biological: Controlled vaccine — The placebo was manufactured by Sinovac Research& Development Co., Ltd.The composition is aluminium hydroxide,The appearance of the placebo is consistent with the vaccine, which is a milky-white suspension.
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
This study is a global multi-center , case-driven, randomized, double-blinded, and placebo-controlled phase Ⅲ clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the efficacy of two dose of CoronaVac® against RT-PCR confirmed symptomatic COVID-19 cases in participants aged 6 months to 17 years.

DETAILED DESCRIPTION:
This study is a global multi-center , case-driven, randomized, double-blinded, and placebo-controlled phase Ⅲ clinical trial in participants aged 6 months to 17 years.The purpose of this study is to evaluate the efficacy of two dose of CoronaVac® against RT-PCR confirmed symptomatic COVID-19 cases in participants aged 6 months to 17 years.The experimental vaccine and placebo were both manufactured by Sinovac Research & Development Co., Ltd. A total of 14,000 healthy participants aged 6 months to 17 years will be enrolled, and randomly assigned into 2 groups at a ratio of 1:1 to receive 2 doses of experimental vaccine (600SU) or placebo with an interval of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adolescents aged 6 months to 17 years;
* The participants and/or their guardians are able to understand and sign the informed consent voluntarily (in accordance with the local regulations);
* Able to comply with study procedures based on the assessment of the Investigator;
* Female participants of childbearing potential (post-menarche girls or in accordance with the local standard of care) may be enrolled in the study if the participant fulfills all the following criteria:

  * Has a negative pregnancy test on the day of the first dose (Day 0).
  * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 0).
  * Has agreed to continue adequate contraception through 3 months following the second dose (Day 28).
  * Is not currently breastfeeding.
* Must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of confirmed infection of SARS CoV-2 prior to randomization;
* Close contact with a confirmed COVID-19 within 14 days prior to randomization;
* Prior administration of an investigational coronavirus vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Allergy to vaccines or vaccine/placebo ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneuroedema;
* Personal or first-grade relative (siblings) history of multisystem inflammatory disease in children (MIS-C);
* Significant chronic illnesses that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion (may include, but are not limited to cardiovascular disease, liver or kidney disorders, respiratory illnesses)
* Significant chronic central nervous system diseases or neuromuscular disorders, psychosis or severe cognitive behavioral disorder, in the opinion of the investigator, including epilepsy, autism spectrum disorder, intellectual disabilities (excluding Down Syndrome);
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* History of autoimmune and/or haematological diseases (including but not limited to systemic lupus erythematosus, thyroidectomy, autoimmune thyroid disease, any form of malignant tumor, asplenia, functional asplenia, or splenectomy resulting from any condition); well controlled type I diabetes mellitus is allowed;
* History of bleeding disorders (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture;
* Immunosuppressive therapy (systemic corticoid therapy, e.g. prednisone ≥2 mg/Kg/d or ≥20 mg/day for >14 days), cytotoxic therapy (antineoplastic chemotherapy, radiation therapy), (excluding topical or aerosol corticosteroid therapy) in the past 6 months;
* Receipt of blood products or immunoglobulins in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc;
* Acute febrile illness with oral temperature >37.7°C or axillary temperature >37.5°C on the day of vaccination (refer to section 7.1 Delay/Discontinuation of Study Vaccination); enrollment could be considered if the fever is absent for 72 hours;
* Any confirmed or suspected human immunodeficiency virus (HIV) infection;
* Children in care or under a court order;
* According to the investigator's judgment, the subject has any other factors that might interfere with the results of the clinical trial or pose additional risk to the subject due to participation in the study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11349 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy index-incidence of RT-PCR confirmed symptomatic COVID-19 cases with onset | 14 days after the second dose
  Incidence of RT-PCR confirmed symptomatic COVID-19 cases with onset at least 14 days after the second dose

SECONDARY OUTCOMES:
Efficacy index-incidence of RT-PCR confirmed symptomatic COVID-19 cases with onset | 14 days after the first dose
  Incidence of RT-PCR confirmed symptomatic COVID-19 cases with onset at least 14 days after the first dose
Efficacy index-incidence of RT-PCR confirmed, symptomatic COVID-19 cases with onset in SARS-CoV-2 uninfected participants | 14 days after the second dose
  Incidence of RT-PCR confirmed, symptomatic COVID-19 with onset at least 14 days after the second dose in SARS-CoV-2 uninfected (serologically or molecularly confirmed) participants at baseline
Efficacy index-incidence of hospitalization/severe/death caused by COVID-19 with onset | 14 days after the second dose
  Incidence of hospitalization/severe/death caused by COVID-19 with onset at least 14 days after the second dose
Safety index-occurrence, intensity, duration, and relationship of solicited local and systemic AEs and of unsolicited AEs | During 7 days following each dose vaccination and during 28 days post-vaccination
  Occurrence, intensity, duration, and relationship of solicited local and systemic AEs during 7 days following each dose vaccination and of unsolicited AEs during 28 days post-vaccination
Safety index-occurrence and relationship of SAEs | From first dose to 12 months after the last dose
  Occurrence and relationship of SAEs from first dose to 12 months after the last dose
Safety index-occurrence and relationship of AESI | From first dose to 12 months after the last dose
  Occurrence and relationship of AESI from first dose to 12 months after the last dose
Immunogenicity index(subgroup)-SARS-CoV-2 neutralizing antibody titers | From first dose to 12 months after the last dose
  Analysis of SARS-CoV-2 neutralizing antibody titers by micro-cytopathic method to compare with the placebo group
Immunogenicity index(subgroup)-Anti-SARS-CoV-2 S | From first dose to 12 months after the last dose
  Analysis of Anti-SARS-CoV-2 S by electrochemiluminescence immunoassay to compare with the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Gang, Doctor, Study Director — Facultad de Medicina, Pontlficla Universidad Católica de Chile
Locations (38):
- Chile (12):
  - Hospital de Puerto Montt, Port Montt, Los Lagos Region
  - Clínica Alemana Valdivia, Valdivia, Los Ríos Region
  - Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Hospital Universidad Clinico de Antofagasta, Antofagasta, Santiago Metropolitan
  - Hospital Roberto del Río, Independencia, Santiago Metropolitan
  - Clínica San Carlos de Apoquindo, Las Condes, Santiago Metropolitan
  - Clínica Universidad de los Andes, Las Condes, Santiago Metropolitan
  - San Joaquín, Macul, Santiago Metropolitan
  - Hospital Sótero del Río, Puente Alto, Santiago Metropolitan
  - Hospital Ezequial Gonzalez, San Miguel, Santiago Metropolitan
  - Marcoleta, Santiago, Santiago Metropolitan
  - Clínica Alemana, Vitacura, Santiago Metropolitan
- Malaysia (10):
  - Hospital Wanita dan Kanak-Kanak Sabah, Kota, Kinabalu Sabah
  - Klinik Kesihatan Cheras Baru, Cheras, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Miri, Miri, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Pengajar UiTM Puncak Alam, Bandar, Selangor
  - Klinik Kesihatan Pandamaran, Port Klang, Selangor
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - University Malaya Medical Centre, Kuala Lumpur
- Philippines (5):
  - Asian Hospital and Medical Center, City of Muntinlupa
  - National Children's Hospital, Manila
  - Philippine Children's Medical Center, Manila
  - Philippine General Hospital, Manila
  - University of Philippines, National Institute of Health, Manila
- South Africa (11):
  - Mecru Clinical Research Unit, Ga-Rankuwa, Gauteng
  - Mecru Clinical Research Unit, Bellville
  - Tiervlei Trial Centre, Bellville
  - Worthwhile Clinical Trials, Benoni
  - Reimed Reicherpark, Boksburg
  - Newtown Clinical Research Centre, Johannesburg
  - Madibeng Centre for Research, Madibeng
  - Be Part Research, Paarl
  - Global Clinical Trials, Pretoria
  - Sandton Medical Research Centre, Sandton
  - Soweto Clinical Trials Center, Soweto

REFERENCES:
- [Derived] Rivera-Perez D, Mendez C, Diethelm-Varela B, Melo-Gonzalez F, Vazquez Y, Meng X, Xin Q, Fasce RA, Fernandez J, Mora J, Ramirez E, Acevedo ML, Valiente-Echeverria F, Soto-Rifo R, Grifoni A, Weiskopf D, Sette A, Astudillo P, Le Corre N, Abarca K, Perret C, Gonzalez PA, Soto JA, Bueno SM, Kalergis AM. Immune responses during COVID-19 breakthrough cases in vaccinated children and adolescents. Front Immunol. 2024 May 15;15:1372193. doi: 10.3389/fimmu.2024.1372193. eCollection 2024. PMID 38812507
- [Derived] Soto JA, Melo-Gonzalez F, Gutierrez-Vera C, Schultz BM, Berrios-Rojas RV, Rivera-Perez D, Pina-Iturbe A, Hoppe-Elsholz G, Duarte LF, Vazquez Y, Moreno-Tapia D, Rios M, Palacios PA, Garcia-Betancourt R, Santibanez A, Pacheco GA, Mendez C, Andrade CA, Silva PH, Diethelm-Varela B, Astudillo P, Calvo M, Cardenas A, Gonzalez M, Goldsack M, Gutierrez V, Potin M, Schilling A, Tapia LI, Twele L, Villena R, Grifoni A, Sette A, Weiskopf D, Fasce RA, Fernandez J, Mora J, Ramirez E, Gaete-Argel A, Acevedo ML, Valiente-Echeverria F, Soto-Rifo R, Retamal-Diaz A, Munoz-Jofre N; PedCoronaVac03CL Study Group,; Meng X, Xin Q, Alarcon-Bustamante E, Gonzalez-Aramundiz JV, Le Corre N, Alvarez-Figueroa MJ, Gonzalez PA, Abarca K, Perret C, Carreno LJ, Bueno SM, Kalergis AM. Inactivated Vaccine-Induced SARS-CoV-2 Variant-Specific Immunity in Children. mBio. 2022 Dec 20;13(6):e0131122. doi: 10.1128/mbio.01311-22. Epub 2022 Nov 16. PMID 36383021